CLINICAL TRIAL: NCT04979637
Title: A Multi Centre, International, Analytical Performance Study of pH, HNE and MPO Levels in Detecting Wound Infection Proof of Concept Biomarker Study
Brief Title: Analytical Performance of pH, HNE and MPO Levels in Detecting Wound Infection Proof of Concept Biomarker Study
Acronym: INDICATE
Status: Withdrawn | Type: Observational
Why Stopped: ConvaTec have been unable to recruit sufficient subjects meeting the inclusion / exclusion criteria and also due to the ongoing Covid-19 restrictions at hospitals and clinics
Sponsor: ConvaTec Inc. (Industry)
Collaborators: ClinSearch (Other); Qualizyme Diagnostics GmbH & Co KG (Industry); Perfectus BioMed (Unknown); Welsh Wound Innovation Centre (Unknown); Maison de Santé Protestante de Bordeaux (Unknown)
Responsible Party: Sponsor
Other Study IDs: WC-20-407
Record Dates: First submitted 2021-07-06; First posted 2021-07-28 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Wound Infection; Wound Heal
Keywords: diabetic foot; pressure ulcer; varicose ulcer
MeSH Terms: conditions — Wound Infection; Diabetic Foot; Pressure Ulcer; Varicose Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a novel combination of biomarkers, pH/HNE/MPO, in detecting wound infection using the clinical judgement at 4 weeks as a standard of reference which will include a wound biopsy.

DETAILED DESCRIPTION:
One of the biggest challenges in wound care today is the accurate and timely diagnosis of infection in complex wounds. Despite efforts, it still remains difficult to determine whether complex wounds are infected or not. There is no single gold standard for wound infection: clinicians use a multitude of methods in addition to the history and their examination to reach an overall conclusion as to potential wound infection status - each with its own strengths and weaknesses (associated performance characteristics).

To aid accurate and timely detection of wound infection in clinical practice, ConvaTec and partners have developed a new technology intended to detect infection biomarkers. This is based on the combined measurement of the following three biomarkers: wound pH, and activity of human neutrophil elastase (HNE) and myeloperoxidase (MPO) host enzymes.

The overall aim of this proof of concept study is to demonstrate that the three infection biomarkers (HNE/MPO/pH) surpass clinical judgement in detecting infection status using a standard of reference.

The primary objective of the proof of concept study is to demonstrate the effectiveness of a novel combination of biomarkers, pH/HNE/MPO, in detecting wound infection using the clinical judgement at 4 weeks as a standard of reference which will include a wound biopsy.

The secondary objective of the proof of concept study is to explore the relationship between molecular microbiological analysis of swab samples and wound biopsies with the biomarkers pH, HNE and MPO.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with an exuding chronic wound, presenting at study sites or associated clinical or home setting
* Aged 18 years and over
* Subjects who are able and willing to provide informed consent.

Exclusion Criteria:

* Subjects with a wound in which it is not possible to take a wound swab:
* Wounds ≤ 2 cm2 in diameter.
* Subjects who are taking or have taken systemic antibiotics in the previous 7 days
* Wounds with scant or no exudate
* Wounds that do not have sufficient exudate to complete swab collection
* Wounds where the wound bed consists predominantly of exposed bone.
* Subjects currently confirmed positive for Methicillin-resistant Staphylococcus aureus (MRSA), extended spectrum beta-lactamase (ESBL) producing bacteria, Human immunodeficiency virus (HIV), hepatitis or severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)
* Subjects on immunosuppressive or cytotoxic drugs
* Anticoagulated patients who cannot undergo wound biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of eligible patients attending their regular wound care appointment with a Health Care Professional in a Clinical setting.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the combination of pH/HNE/MPO, in detecting wound infection using the clinical judgement at 4 weeks as a standard of reference which will include a wound biopsy | Day 28
  This will be expressed as the diagnostic properties: positive and negative predictive values, and area under the receiver operating characteristic curve, for the three markers alone and in different combinations.

SECONDARY OUTCOMES:
Explore the relationship between molecular microbiological analysis of swab samples and wound biopsies with the biomarkers pH, HNE and MPO. | Day 28
  Data obtained from the study will be analysed in order to further understand the relationship between molecular microbiological analysis of swab samples and wound biopsies with the biomarkers pH, HNE and MPO.

CONTACTS AND LOCATIONS:
Overall Officials: Nicky Irvins, Principal Investigator — Welsh Wound Innovation Centre